CLINICAL TRIAL: NCT03876574
Title: Hepatic Artery Infusion Gemcitabine and Floxuridine in Patients With Nasopharyngeal Carcinoma Liver Metastases
Brief Title: Hepatic Artery Infusion Pump for NPC Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC11330
Record Dates: First submitted 2019-03-03; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Nasopharyngeal Carcinoma; Neoplasm Metastasis; Liver
Keywords: Hepatic artery infusion pump; Gemcitabine; Floxuridine
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — Gemcitabine; Floxuridine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients undergo DSA-guided implantation of hepatic artery infusion pump. All patients receive the intervention "Hepatic artery infusion of gemcitabine and floxuridine" the next day after pump implantation. The HAI therapy is initiated on day 1, 8: Gemcitabine 1g/m2 for 30 minutes, followed by a blended solution which comprised floxuridine (FUDR) at 0.15 mg/kg/day, dexa-methasone (DXM) at 1 mg/m2/day, low molecular heparin 3200U and saline, lasted for 7 days continuously.Standard treatments of NPC, including radiotherapy and chemotherapy (induction chemotherapy, concurrent chemotherapy and adjuvant chemotherapy) are performed as desired.
  Interventions: Procedure: DSA-guided implantation of hepatic artery infusion pump; Drug: Gemcitabine; Drug: Floxuridine; Drug: dexamethasone

INTERVENTIONS:
Procedure: DSA-guided implantation of hepatic artery infusion pump — Implant the infusion catheter and injection port (Celsite, B. Braun, Chasseneuil, France) under DSA-guiding. The proximal end of the infusion catheter was connected to the injection port and the device was implanted in a subcutaneous pocket in the right inner thigh; the distal end of the infusion catheter guarantee uni-direction infusion to liver.
Drug: Gemcitabine — Given intra-arterially for 30 minutes
Drug: Floxuridine — Given intra-arterially continuously for 14 days
  Other Names: 5-FUDR
Drug: dexamethasone — Given intra-arterially continuously with 5-FUDR
  Other Names: DXM

SUMMARY:
A retrospective clinical trial to study the safety and effectiveness of hepatic arterial infusion (HAI) in treating patients who have nasopharyngeal carcinoma metastatic to the liver. Hepatic-direction drug administration improves the control power for intra-hapatic lesions.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety and toxicity of hepatic arterial infusion with gemcitabine, floxuridine and dexamethasone in combination with standard treatment (radiotherapy and systemic chemotherapy) in patients with nasopharyngeal carcinoma metastases to liver.

II. Determine the objective response of intrahepatic lesions of patients treated with this regimen.

III. Determine the median survival time or overall survival time in patients treated with this regimen.

OUTLINE: This is a single-center retrospective study.

Patients receive DSA-guided implantation of HAI catheter system. HAI is initiated the next day. Gemcitabine intra-arterially for 30 minutes on day 1,8, floxuridine, dexamethasone intra-arterially continuously on days 1-14. Treatment repeats every 3 weeks in the absence of serious technical catheter-related problems, progression of intrahepatic lesions or unacceptable toxicity. Standard treatment of NPC, including radiotherapy and chemotherapy (induction chemotherapy, concurrent chemotherapy and adjuvant chemotherapy) was performed as desired.

Patients are followed every 2 HAI cycles or when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed nasopharyngeal carcinoma with histologically confirmed or image diagnosed metastatic to the liver
* Standard treatment of NPC, including radiotherapy and chemotherapy (induction chemotherapy, concurrent chemotherapy and adjuvant chemotherapy) is performed as desired
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* No pre-existing chronic hepatic disease (chronic active hepatitis or cirrhosis)
* Creatinine no greater than ULN
* Creatinine clearance greater than 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate oral nutrition (at least 1,500 calories/day)
* Able to withstand major operative procedure
* No dehydration
* No severe anorexia
* No frequent nausea or vomiting
* No prior or concurrent malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of any organ
* No prior or concurrent malignancy associated with more than 10% probability of death from malignant disease within 5 years of diagnosis
* No concurrent immunotherapy
* No concurrent colony-stimulating factors during the first course of study therapy
* No more than 1 prior adjuvant systemic fluorouracil (5-FU) regimen with or without levamisole, leucovorin calcium, or irinotecan
* No prior hepatic artery infusion therapy with 5-FU or floxuridine
* No prior systemic chemotherapy for metastatic disease
* No prior or concurrent sorivudine or brivudine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) of intrahepatic lesions | 2 years
  Assess the Disease control rate (DCR) of intrahepatic lesions by enhanced spiral-CT scan according to RECIST criteria.

SECONDARY OUTCOMES:
Overall survival time | 7 years
  From the date of HAI catheter implantation to the date of death from any cause or to completion of trial, whichever comes first, up to 84 months.
Side effects and adverse events | 2 years
  To determine the safety and tolerability of HAI for NPC liver metastases by establishing the rates of toxicity